CLINICAL TRIAL: NCT00505440
Title: Trial of Automated Risk Appraisal for Adolescents
Acronym: TARAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelly Kelleher, Professor of Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 5R01DA018943-04 (NIH); R01DA018943 (NIH)
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Substance Use; Depression; Suicidal Ideation; Risk Behavior
MeSH Terms: conditions — Substance-Related Disorders; Depression; Suicidal Ideation; Risk-Taking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized screening and referral (Experimental): Computerized screening and referral: Intervention is a web-based screening and assessment tool completed by adolescents during primary care visits. Patient reported screening provided to primary care physicians in real time with recommendations for behavioral referrals.
  Interventions: Behavioral: Telephone case management and motivational interviewing
- Delayed feedback from screening (Active Comparator): Active comparator is Usual pediatric care plus mailed screening results from computerized waiting room screens that arrive three days after screening.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Telephone case management and motivational interviewing — 'Telephone case management and motivational interviewing': Immediate screening results are given to the physician during the patient's visit. Telephone case management and motivational interviewing (MI) at 1, 6, and 9 weeks to enhance engagement and commitment to change
  Arms: Computerized screening and referral
Behavioral: Usual care — Usual care with mailed screening results
  Arms: Delayed feedback from screening

SUMMARY:
This is a study to find out which type of computer screening and nursing support can improve screening for high risk behaviors in doctor's offices. Recommendations call for doctors to screen young people for many different behaviors and feelings such as depression, not wearing seat belts, alcohol and drug use. Doctors rarely have time to complete these screenings. New computers can help ask some of these questions and protect patient information. In addition, nurse telephone calls can often help young persons with some of the behaviors receive treatment. This study will examine which type of computer screening and follow-up will help patients the most.

DETAILED DESCRIPTION:
The pandemic of problem drug use and abuse and related health problems among young persons aged 12-25 in the U.S. continues unabated, in part, because opportunities for early identification and monitoring are missed. In particular, improved recognition of, and ongoing contact for, problem drug use and abuse among pre-teens and early adolescents in primary care settings could provide important information to health care professionals and engage early intervention services. Unfortunately, many barriers exist to routine screening and monitoring in primary care settings. These include the expense of traditional paper and pencil screening, competing demands on primary care clinicians and office staff, complex scoring programs and the ability to track youth over time.

Innovative information technology and support services can overcome many of these barriers. New primary care information systems allow for direct data entry by youth in healthcare settings, automated scoring and printing, decreased staff time, individual or practice level results and patient follow-up for intervention services. However, these assessment tools and systems have not been adequately assessed for their roles in detecting problem drug use and abuse in youth, and appropriate follow-up and tracking systems for those identified have not been implemented.

Our goal is to improve services for problem drug use and abuse and other related health risking behaviors for youth in primary care settings through early identification and monitoring. We expand an innovative partnership among the Columbus Children's Hospital, the Close To Home Primary Care Centers and Flipsidemedia.com to test the efficacy and acceptability of an early identification and monitoring system for problem drug use and abuse, depression and related mental disorders among pre-teens and teenagers in a randomized trial. We propose to compare care in nine Close To Home Centers with Automated Risk Appraisal for Adolescents/Telephone Support (RA/TS) compared to usual care plus mailed screening results (UC+). Each site will be randomly assigned to start with six months on RA/TS or six months on UC+ and follow with the alternative in a crossover design. RA/TS is a web-based screening and assessment tool completed by adolescents during primary care visits and a linked, structured telephone tracking intervention consisting of three follow-up telephone calls to youth and their families monitoring identified problems and barriers to services. Specifically, we aim to:

1. compare frequency of problem drug use and abuse identification in RA/TS youth vs. youth in usual care (UC+);
2. examine frequency of counseling, referral, psychotropic medication or other interventions for youth screening positive for problem drug use and abuse on RA (Risk Appraisal) in RA/TS youth vs. UC+ youth; and
3. evaluate the effects of the TS (Telephone Support) program on return to primary care, likelihood of completing referrals, number of primary care visits, number of specialty visits, and satisfaction with services after four months for youth screening positive for problem drug use and abuse.

ELIGIBILITY:
Inclusion Criteria:

* 11-20 years of age
* non-emergent visit in primary care office
* consent and assent (if applicable)

Exclusion Criteria:

* non-english speaking

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1185 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
identification of problem drug use and abuse, depression, and other mental disorders using the Automated Risk Appraisal for Adolescents / Telephone Support (RA/TS) tool compared with usual care practices | 6 months

SECONDARY OUTCOMES:
receipt of counseling services | 6 months
referral to mental health and other services | 6 months
medications for mental health disorders | 6 months
return to primary care | 6 months
completion of referrals | 6 months
number of primary care visits | 6 months
number of specialty visits | 6 months
satisfaction with RA/TS services | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Kelleher, MD, MPH, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Columbus Children's Research Institute, Columbus, Ohio, United States

REFERENCES:
- [Background] Penfold RB, Kelleher KJ. Use of surveillance data in developing geographic dissemination strategies: a study of the diffusion of olanzapine to Michigan children insured by medicaid. Clin Ther. 2007 Feb;29(2):359-70; discussion 358. doi: 10.1016/j.clinthera.2007.02.017. PMID 17472829
- [Background] Julian TW, Kelleher K, Julian DA, Chisolm D. Using technology to enhance prevention services for children in primary care. J Prim Prev. 2007 Mar;28(2):155-65. doi: 10.1007/s10935-007-0086-8. Epub 2007 Feb 6. PMID 17279327
- [Background] Kaizar E, Chisolm D, Seltman H, Greenhouse J, Kelleher KJ. The role of care location in diagnosis and treatment of pediatric psychosocial conditions. J Dev Behav Pediatr. 2006 Jun;27(3):219-25. doi: 10.1097/00004703-200606000-00007. PMID 16775519
- [Background] Gardner W, Shear K, Kelleher KJ, Pajer KA, Mammen O, Buysse D, Frank E. Computerized adaptive measurement of depression: a simulation study. BMC Psychiatry. 2004 May 6;4:13. doi: 10.1186/1471-244X-4-13. PMID 15132755
- [Background] Gardner W, Kelleher KJ, Pajer KA. Multidimensional adaptive testing for mental health problems in primary care. Med Care. 2002 Sep;40(9):812-23. doi: 10.1097/00005650-200209000-00010. PMID 12218771
- [Background] Chisolm DJ, Young RR, McAlearney AS. Implementation of a touch-screen new patient registration system: a case study. J Med Pract Manage. 2005 Nov-Dec;21(3):159-62. PMID 16471390
- [Derived] Stevens J, Kelleher KJ, Gardner W, Chisolm D, McGeehan J, Pajer K, Buchanan L. Trial of computerized screening for adolescent behavioral concerns. Pediatrics. 2008 Jun;121(6):1099-105. doi: 10.1542/peds.2007-1878. PMID 18519478